CLINICAL TRIAL: NCT04323072
Title: Influence of the Size of the Gastric Antrum After Sleeve Gastrectomy on Weight Loss in Bariatric Surgery
Brief Title: Does Antrum Size Matter in Sleeve Gastrectomy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Head of the bariatric and metabolic surgery unit, Azienda Sanitaria Locale Napoli 2 Nord
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01032020
Record Dates: First submitted 2020-03-18; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Resection of antrum proximally 2 cm to the pylorus
  Interventions: Procedure: Wide antrectomy
- Group B (Active Comparator): Resection of antrum proximally 6 cm to the pylorus
  Interventions: Procedure: Smal antrectomy

INTERVENTIONS:
Procedure: Wide antrectomy — The starting point of resection of the stomach from the pylorus to begin the gastrectomy is 2 cm.
  Arms: Group A
Procedure: Smal antrectomy — The starting point of resection of the stomach from the pylorus to begin the gastrectomy is 6 cm.
  Arms: Group B

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) is currently the most frequent primary bariatric procedure performed worldwide. LSG is safe and effective in terms of excess weight loss. It is a powerful metabolic operation that activates significant hormonal pathways that lead to changes in eating behaviour, glycemic control and intestinal functions. LSG is easier regarding its technical aspects and does not need any intestinal anastomosis, begin limited to the stomach. The most frequent and sometimes dangerous complications are leaking, haemorrhage, splenic injury, sleeve stenosis and gastroesophageal reflux. Despite its established efficacy and safety, controversy still exists on optimal operative technique for LSG: bougie size, the distance of resection margin from the pylorus, the shape of the section at the gastroesophageal junction, staple line reinforcement and intraoperative leak testing is among the most controversial issues 11[6]. In literature, different authors have adopted a resection distance from the pylorus between 2 and 6-7 cm with various reasons 11[6]. Resections more distant to the pylorus improve gastric emptying, prevent distal stenosis and reduce intraluminal pressure, potentially leading to a lower incidence of fistula and/or reflux. On the other hand, resections close to the pylorus would reduce gastric distensibility and increase intragastric pressure, potentially increasing satiety with less oral intake 11(11,12). The primary aim of this randomized monocentric study is to evaluate %EWL at 1 and 2 years follow-up after LSG in two Groups: Group A with a gastric resection starting from 2 cm from the pylorus with therefore a wide antrectomy and Group B with a gastric resection starting from 6 cm from the pylorus with therefore a small antrectomy.

ELIGIBILITY:
Inclusion criteria:

* informed consent.
* morbid obesity defined as body mass index (BMI) 40 kg/m2

Exclusion Criteria:

* previous bariatric surgical procedures,
* endocrine disorders causing obesity
* pregnancy or lactation
* psychiatric illness
* inflammatory bowel disease
* Barrett ́s oesophagus
* severe GERD with esophagitis B and C
* a large hiatal hernia (>5 cm)
* GERD-HRQLscore > 25 dietary restriction despite

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative weight and height combined to report BMI in kg/m^2 | 3 months
  Change of weight and height expressed in Postoperative Body Mass Index obtained by dividing the weight by the squared height expressed in meters (kg/m2)
Postoperative weight and height combined to report BMI in kg/m^2 | 6 months
  Change of weight and height expressed in Postoperative Body Mass Index obtained by dividing the weight by the squared height expressed in meters (kg/m2)
Postoperative weight and height combined to report BMI in kg/m^2 | 12 months
  Change of weight and height expressed in Postoperative Body Mass Index obtained by dividing the weight by the squared height expressed in meters (kg/m2)
Postoperative weight and height combined to report BMI in kg/m^2 | 24 months
  Change of weight and height expressed in Postoperative Body Mass Index obtained by dividing the weight by the squared height expressed in meters (kg/m2)
Postoperative percentage excess weigth loss | 3 months
  Change of weight expressed in percentage of excess weight loss postoperatively at follow-up
Postoperative percentage excess weigth loss | 6 months
  Change of weight expressed in percentage of excess weight loss postoperatively at follow-up
Postoperative percentage excess weigth loss | 12 months
  Change of weight expressed in percentage of excess weight loss postoperatively at follow-up
Postoperative percentage excess weigth loss | 24 months
  Change of weight expressed in percentage of excess weight loss postoperatively at follow-up

SECONDARY OUTCOMES:
Gastroesophageal reflux disease(GERD) | at 12 months
  Esophagitys grading according to Los Angeles classification with Upper endoscopy (Grade A: One or more mucosal breaks < 5 mm in maximal length; Grade B: One or more mucosal breaks > 5mm, but without continuity across mucosal folds; Grade C: Mucosal breaks continuous between ≥ 2 mucosal folds, but involving less than 75% of the esophageal circumference Grade D Mucosal breaks involving more than 75% of esophageal circumference
Gastroesophageal reflux disease(GERD) | at 24 months
  Esophagitys grading according to Los Angeles classification with Upper endoscopy (Grade A: One or more mucosal breaks < 5 mm in maximal length; Grade B: One or more mucosal breaks > 5mm, but without continuity across mucosal folds; Grade C: Mucosal breaks continuous between ≥ 2 mucosal folds, but involving less than 75% of the esophageal circumference Grade D Mucosal breaks involving more than 75% of esophageal circumference
Gastroesophageal reflux disease symptoms | at 3 months
  All patients were surveyed about the presence of heartburn and/or regurgitation with a specific questionnaire GERD HRQL(Gastroesophageal Reflux Disease Health-Related Quality of Life) questionnaire. Each of the 10 questions were rated from 0 (absence of symptoms) to 5 (severe symptoms) for a total score that may range from 0 to 50. Symptoms were defined as absent when patients reported a GERD-HRQL score of 0, mild from 1 to 15, moderate from 16 to 24, and severe from 25 to 50.
  Patients with GERD-HRQL score >16 was considered positive for GERD.
Gastroesophageal reflux disease symptoms | at 6 months
  All patients were surveyed about the presence of heartburn and/or regurgitation with a specific questionnaire GERD HRQL(Gastroesophageal Reflux Disease Health-Related Quality of Life) questionnaire. Each of the 10 questions were rated from 0 (absence of symptoms) to 5 (severe symptoms) for a total score that may range from 0 to 50. Symptoms were defined as absent when patients reported a GERD-HRQL score of 0, mild from 1 to 15, moderate from 16 to 24, and severe from 25 to 50.
  Patients with GERD-HRQL score >16 was considered positive for GERD.
Gastroesophageal reflux disease symptoms | at 12 months
  All patients were surveyed about the presence of heartburn and/or regurgitation with a specific questionnaire GERD HRQL(Gastroesophageal Reflux Disease Health-Related Quality of Life) questionnaire. Each of the 10 questions were rated from 0 (absence of symptoms) to 5 (severe symptoms) for a total score that may range from 0 to 50. Symptoms were defined as absent when patients reported a GERD-HRQL score of 0, mild from 1 to 15, moderate from 16 to 24, and severe from 25 to 50.
  Patients with GERD-HRQL score >16 was considered positive for GERD.
Gastroesophageal reflux disease symptoms | at 24 months
  All patients were surveyed about the presence of heartburn and/or regurgitation with a specific questionnaire GERD HRQL(Gastroesophageal Reflux Disease Health-Related Quality of Life) questionnaire. Each of the 10 questions were rated from 0 (absence of symptoms) to 5 (severe symptoms) for a total score that may range from 0 to 50. Symptoms were defined as absent when patients reported a GERD-HRQL score of 0, mild from 1 to 15, moderate from 16 to 24, and severe from 25 to 50.
  Patients with GERD-HRQL score >16 was considered positive for GERD.

CONTACTS AND LOCATIONS:
Locations (1):
- Francdesco Pizza, Napoli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT04323072/Prot_SAP_000.pdf